CLINICAL TRIAL: NCT01834118
Title: Reintervention After Previous Renal Denervation in Non-responding Patients With Severe Hypertension
Brief Title: Reintervention-study After Previous Renal Denervation in Non-responding Patients With Severe Hypertension
Acronym: RETREAT
Status: Completed | Type: Observational
Sponsor: Cardiovascular Center Frankfurt (Other)
Responsible Party: Principal Investigator, Prof. Dr. Horst Sievert, M.D., Cardiovascular Center Frankfurt
Other Study IDs: CVC-001
Record Dates: First submitted 2013-04-15; First posted 2013-04-17 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Hypertension, Resistant to Conventional Therapy
MeSH Terms: conditions — Hypertension Resistant to Conventional Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Renal Denervation — Sympathetic nerve ablation via transcatheter renal denervation
  Other Names: Renal sympathetic nerve ablation

SUMMARY:
The purpose of this study is to determine the effect of repeated renal denervation in non-responding patients with severe hypertension. Therefore ultrasound technique will be used.

DETAILED DESCRIPTION:
Renal Denervation is a CE-certified opportunity for treating patients with therapy-refractory hypertension. In some patients it doesn't show a significant lowering of the blood pressure, so a repeated renal denervation is an option.

In this study repeated renal denervation will be performed with the Recor Paradise Ultrasound Catheter.

For the study no specific procedures are required which would exceed the standard renal denervation procedure with the CE-certified Recor Paradise Ultrasound Catheter System.

There are no additional risks for the patient in consequence of participating in the study or the follow up procedures.

ELIGIBILITY:
Inclusion Criteria:

* Individual is ≥18 years old
* Individual received renal denervation ≥12 months prior to study participation to no therapeutical avail and is scheduled for reintervention.
* Systolic Office based blood pressure ≥140mmHg
* Individual receives 3 or more antihypertensive drugs including one diuretic
* Individual is willing to provide written informed consent to participate in this study

Exclusion Criteria:

* Individual has hypertension secondary to an identifiable and treatable cause
* Individual has any serious medical condition which in the opinion of the investigator may adversely affect the participation.
* Individual is pregnant, nursing or planning to be pregnant
* Renal artery abnormalities which may affect the procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with treatment-resistant hypertension, who already underwent renal denervation with no therapeutic avail.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2013-06; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Office Blood pressure measurement | up to1 year

CONTACTS AND LOCATIONS:
Overall Officials: Horst Sievert, M.D., Principal Investigator — Cardiovascular Center Frankfurt
Locations (1):
- CardioVascular Center Frankfurt, Frankfurt am Main, Hesse, Germany